CLINICAL TRIAL: NCT00812474
Title: Regional Cortical Cerebral Quantitative MRI Perfusion Correlation Neurocognition in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Unity Health Toronto (Other); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dr. Richard Aviv, PI, Sunnybrook Health Sciences Centre
Other Study IDs: 373-2007
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Sclerosis
Keywords: cerebral blood flow
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multiple Sclerosis (MS) is a common disease affecting 1/1000 Canadians. Cognition impairment is reported in 40-65% of patients and is socially and functionally disabling. Although multiple sclerosis is widely regarded as a white matter disease, cortical disease burden is increasingly emphasized. Studies confirm that gray matter (GM) disease is grossly underestimated by conventional MRI. Although the cause for MS is unknown vascular impairment is implicated in nerve cell death. Several studies have shown perfusion abnormalities in the central GM and white matter (WM) structure. Severity of perfusion reduction correlates with lesion load, atrophy, MS subtype and disease duration. Further extent of cortical atrophy correlates with neurocognitive impairment. We hypothesize that cortical perfusion is a marker of cortical disease severity and correlates with neurocognitive impairment. To show this we will measure regional cortical perfusion and regional brain and WM lesion volumes in 26 predefined brain regions using a template developed for Alzheimer's disease. Regional perfusion will be correlated with neurocognitive tests validated for MS use. Patients will be divided into impaired and non impaired and perfusion compared controlling for known confounding factors. If confirmed cortical perfusion may be utilized as a surrogate marker of cognitive outcome in therapeutic studies.

DETAILED DESCRIPTION:
We hypothesize that cortical perfusion is a marker of cortical disease severity and correlates with neurocognitive impairment. To show this we will measure regional cortical perfusion and regional brain and WM lesion volumes in 26 predefined brain regions using a template developed for Alzheimer's disease. Regional perfusion will be correlated with neurocognitive tests validated for MS use. Patients will be divided into impaired and non impaired and perfusion compared controlling for known confounding factors. If confirmed cortical perfusion may be utilized as a surrogate marker of cognitive outcome in therapeutic studies.

ELIGIBILITY:
Inclusion Criteria:

* established SPMS according to the McDonald criteria

Exclusion Criteria:

* Patients with a history of drug/alcohol abuse, a premorbid (pre MS) psychiatric history, a head injury with loss of consciousness and a concurrent physical disease requiring medical attention (eg. cardiovascular disease etc), MRI contraindication including implants, pacemaker, aneurysm clips and known renal impairment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Secondary progressive Multiple sclerosis
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Cognitive Impairment | Cognitive impairment is assessed on the same day as the MRI scan